CLINICAL TRIAL: NCT06477939
Title: Phase III Randomized Study of Adding or Not Liposomal Transcrocetin (L-TC) With Concomitant HypoFractionated Radiation ThErapy and TEmozolomide in Newly Diagnosed GLioblastoma (GBM) Patients to Evaluate Efficacy and Safety
Brief Title: Study of Adding or Not Liposomal Transcrocetin (L-TC) With Concomitant HypoFractionated Radiation ThErapy and TEmozolomide in Newly Diagnosed GLioblastoma (GBM) Patients
Acronym: THREE-GLEES
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: LEAF4Life, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-008; 2024-515666-13-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Glioblastoma
Keywords: Brain tumors; Hypoxia; Liposomal transcrocetin
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Hypoxia | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Radiotherapy plus Temozolomide (Active Comparator)
  Interventions: Drug: Administration of L-TC
- Administration of L-TC on top of Radiotherapy plus Temozolomide (Experimental)
  Interventions: Other: Radiotherapy plus Temozolomide

INTERVENTIONS:
Drug: Administration of L-TC — Administration of L-TC (300 mg) as an IV perfusion, before each radiotion session
  Radiotherapy : delivered at 40.5 Gy in 15 fractions of 2.7 Gy - One fraction a day 5 fractions per week
  + Temozolomide delivered at a dose of 75 mg per square meter per day, given 7 days per week from the first day of radiotherapy until the last day of radiotherapy, but for no longer than 25 days.
  Arms: Radiotherapy plus Temozolomide
Other: Radiotherapy plus Temozolomide — Radiotherapy : delivered at 40.5 Gy in 15 fractions of 2.7 Gy - One fraction a day 5 fractions per week
  + Temozolomide delivered at a dose of 75 mg per square meter per day, given 7 days per week from the first day of radiotherapy until the last day of radiotherapy, but for no longer than 25 days.
  Arms: Administration of L-TC on top of Radiotherapy plus Temozolomide

SUMMARY:
This is phase III randomized, multicenter study adding or not intra-venous Liposomal Trasncrocetin (L-TC) to hypofractionated radiotherapy and concomitant Temozolomide followed by adjuvant Temozolomide in patients with histologically confirmed diagnosis of glioblastoma (GBM).

DETAILED DESCRIPTION:
During this trial the L-TC will be administered with the hypofractionated chemoradiation treatment to two cohorts:

* Cohort 1 - Non-operable population defined as patients with age less than 70-year-old and with biopsy alone, Karnofski index we propose to use the L-TC with the hypofractionated chemoradiation treatment to two cohorts:
* Cohort 2 - Elderly population defined as patients aged of more than 70-year-old and with Balducci score 1 or with low Balducci score 2 with Karnofski index ≥ 70% but whatever the quality of the surgery. For patients classified with a score of Balducci II, the geriatric assessment is essential. Although we are aware of the heterogeneity of patients in this group, we hope that the geriatric assessment will make it possible to reduce this heterogeneity by including only patients with a Charlson score <4 and a score of autonomy IADL = 4

The eligible population will be randomized this combination with the treatment reference according to Perry et al publication

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 - Non-operable patients

  * Patients aged at least 18 years old and ≤ 70 years old; male or female.
  * AND available biopsy
  * AND Karnofsky index ≥ 50% at Screening
* Cohort 2 - Elderly patients

  * Patients aged > 70 years old; male or female
  * AND Balducci score I or II. For patients classified in Balducci II, only light Balducci II will be included, as defined by a Charlson score <4 and a score of autonomy IADL = 4. In the oncogeriatric evaluation, symptoms related to brain cancer disease have not to be considered for this criterion.
  * Karnofsky score (KPS) of ≥ 70% at Screening
  * Regardless resection
  * MRI at maximum 48h00 after surgery if partial, subtotal or macroscopically complete or supra-total resection
* For both cohorts

  * Histologically confirmed diagnosis of glioblastoma (GBM) (2016 OMS classification) (Louis et al., 2016).
  * Contrast enhancing disease on MRI within 14 days prior to screening.
  * Within 2 weeks of baseline visit, hematologic and renal functions as specified: Absolute neutrophil count ≥ 1500/mm3, platelets ≥ 100,000/mm3, Hgb ≥ 9.0g/dL, creatinine ≤ 1.7mg/dl, total bilirubin ≤ 1.5mg/dL, blood urea nitrogen (BUN) within 2 times the upper limit of normal, transaminases ≤ 4 times above the upper limits of the institutional norm.
  * Sexually active patients must use an acceptable method of contraception while receiving doses of study medication.
  * Females of childbearing potential must have a negative serum or urine pregnancy test at screening and have additional pregnancy tests during study.

Exclusion Criteria:

• For both cohorts

* Any previous radiotherapy (RT) of the brain whatever the interval between previous brain RT and diagnoses of GBM)
* Any previous treatment of the GBM (except surgery) such as chemotherapy (including Gliadel wafer or gliasite application), immunotherapy, therapy with a biologic agent, hormonal therapy or Carmustine implant for brain tumors or immunotherapy, including vaccination (whatever the interval between previous treatment and diagnoses of GBM). Glucocorticoid therapy is allowed.
* Previous digestive disease with mis-absorption such as Crohn disease or chronic colitis
* Ongoing diarrhea grade ≥ 2 in the NCI CTCAE V5.0 (whatever the cause)
* Inclusion in another trial in the 30 previous days
* Patient who cannot undergo MRI
* Pregnant or lactating woman.
* Serious concurrent infection or medical illness that would jeopardize the ability of the patient to receive study treatment with reasonable safety.
* Patients with previous cancer (< 5 years) except basocellular skin tumors and in situ cervix tumor
* Patient has a known hypersensitivity to crocetins, L-TC or any of its excipients.
* Contraindication of temozolomide as described in the Summary of product characteristics.
* Patient who cannot understand French language.
* Patient without French National Health insurance
* Patient who cannot be reliable for follow-up
* Patient under law protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 24 months
  Overall Survival (OS) is defined as the length of time from the date of tumor resection surgery or definitive biopsy to the date of death.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months
  RANO criteria will be used to evaluate response
Evaluation of hypoxia markers | Up to 24 months
  Hypoxia imaging markers between two groups: comparison of volumetric metrics
Quality of life | Up to 24 months
  European Organisation for Research and Treatment of Cancer (EORTC) 30-Item Core Quality of Life Questionnaire (QLQ-C30)
Quality of life (GBM module) | Up to 24 months
  EORTC 20-Item QOL-Brain Neoplasm (QLQ-BN20)
Quality of life (specific for elderly population) | Up to 24 months
  Quality-of-Life Questionnaire EORTC Elderly Cancer Patients (EORTC QLQ-ELD14)
Tolerance | Up to 24 months
  EORTC Elderly Cancer Patients (EORTC QLQ-ELD14)

CONTACTS AND LOCATIONS:
Overall Officials: Georges NOEL, MD, PhD, Principal Investigator — Institut de cancérologie Strasbourg Europe
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France